CLINICAL TRIAL: NCT05587920
Title: The Effect of Menstrual Cycle Phase and Hormonal Contraceptives on Bone Metabolism, Reproductive Status, Iron Status and Musculoskeletal Health
Brief Title: Effect of Oestrogen on Musculoskeletal Outcomes
Acronym: E2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Army Health Branch, British Army (Other Government)
Collaborators: University of East Anglia, Norwich, United Kingdom (Unknown); Osteolabs, Kiel, Germany (Unknown); University of Salford, Salford, United Kingdom (Unknown); University of Southampton, Southampton, United Kingdom (Unknown)
Responsible Party: Principal Investigator, Dr. Thomas O'Leary, Higher Scientific Officer, Army Health Branch, British Army
Other Study IDs: 1042/MODREC/20
Record Dates: First submitted 2022-09-02; First posted 2022-10-20 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Contraception; Estrogen Deficiency; Estrogen Excess

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Non-hormonal contraceptive users: Women not using any form of hormonal contraceptive.
- Combined oral contraceptive pill users: Women using the oral combined oral contraceptive pill.
- Hormonal IUS: Women using the hormonal intrauterine system contraceptive.
- Hormonal implant: Women using the hormonal contraceptive implant contraceptive.
- Hormonal injection: Women using the hormonal injection contraceptive.

SUMMARY:
This cross-sectional comparison and prospective cohort design study will investigate differences in calcium metabolism, biochemical markers of bone and reproductive health, musculoskeletal health, and iron status between women using different hormonal contraceptives (combined oral contraceptive pill (COCP), hormonal implant, hormonal intra-uterine system (IUS), hormonal contraceptive injection, and eumenorrheic non-hormonal contraceptive users). The same outcomes will also be examined across a menstrual cycle in the eumenorrheic non-hormonal contraceptive users.

The study will test the following hypotheses:

Hormonal contraceptive use

1. Biochemical markers of bone resorption and formation and ratio of urinary 44Ca:42Ca will be higher in the implant and injection groups compared with IUS (which exerts localised effects) and non-HC users (ovulatory phase), and lower in COCP compared with non-HC users;
2. Oestradiol and progesterone will be lower in hormonal contraceptive users compared with non-HC users during the ovulatory phase;
3. Bone macro- and microstructure, muscle strength, and tissue properties are different in hormonal contraceptive users compared with non-HC users;
4. Calcium and bone metabolism, reproductive hormones and musculoskeletal function are different between the pill phase and non-pill phase of COCP use.

Menstrual cycle phase

1. Calcium and bone metabolism are lower during the ovulatory phase compared with menses, mid follicular and mid luteal phases.
2. Muscle strength and tissue properties are different across the menstrual cycle in non-HC users.

DETAILED DESCRIPTION:
Women of reproductive age experience cyclical variation during the menstrual cycle in the female sex steroid hormones, oestrogens and progesterone. Oestrogens performs a primary function in sexual development and reproduction; but, non-reproductive effects on bone, muscle, sinew tissue (e.g. ligaments and tendons) and metabolism may influence injury risk and physical performance. Hormonal contraceptive use, which is common in athletes and military service women, disrupts the reproductive axis and suppresses endogenous hormone production. The purpose of this study is to compare calcium metabolism, biochemical markers of bone and reproductive health, iron status and musculoskeletal health between women using one of four methods of hormonal contraceptives-combined oral contraceptive pill (COCP), hormonal implant, hormonal intra-uterine system (IUS) and hormonal contraceptive injection-and eumenorrheic, non-hormonal contraceptive users (non-HC).

The study will involve a pre-screening visit followed by the main study visits. During the pre-screen visit a venous blood sample will be taken to assess vitamin D status alongside several questionnaires to evaluate health and lifestyle and determine eligibility. Eumenorrheic women will be given a commercially available fertility tracking wearable bracelet (Ava Science Inc.) which will be worn throughout at least two menstrual cycles in the non-HC group for prediction and detection of ovulation. Following pre-screen, the non-HC group will attend the laboratory on four occasions corresponding to the start of the menstrual bleed, the mid-follicular phase, ovulatory phase and mid-luteal phase; the COCP users will attend on two occasions corresponding to the end of the pill phase and the end of the pill-free phase; and the Long Acting Reversible Contraceptives (LARC) users (hormonal injection, hormonal implant, IUS) will attend for a single study visit. On each study visit, participants will provide a urine and venous blood sample, undertake muscle function tests (isokinetic dynamometry and single-leg drop) and have tendon, muscle and ligament characteristic measurements taken (digital palpation). Bone measurements (DXA, HRpQCT, ultrasound) will be taken on one occasion, (day 14 for the non-HC group; day 21 for the COCP group (i.e. end of pill-using weeks); and the single testing day for other LARC groups. The final measurement of impact microindentation (IMI) will be performed using the Osteoprobe within 4 weeks after the skeletal imaging; the IMI is a specialised procedure and will be scheduled in set sessions each month.

Primary Outcomes: Bone calcium balance (44Ca:42Ca) measured in urine.

Secondary Outcomes: Markers of bone turnover, reproductive function, iron status and musculoskeletal health.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-40 years old
2. No hormonal contraceptive use (with regular menstrual cycles 24-35 days in length, and have not been taking any hormonal contraceptives for at least 12 months), or;
3. Use of the combined oral contraceptive pill containing ≥25 mg ethinyl-oestradiol (EE) and an anti/low androgenic progestin for at least 12 months, or;
4. Use of the hormonal coil (IUS) continuously for at least 2 years, or;
5. Use of the hormonal implant continuously for at least 2 years, or;
6. Use of the hormonalDMPA injection continuously for at least 2 years;
7. Weight stable (no change in self-reported body mass ≥ 5% over the previous 3 months);
8. BMI between 18 and 30 kg·m2.

Exclusion Criteria:

1. Taking a hormonal contraceptive other than the combined oral contraceptive pill containing ≥25 mg EE and an anti/low androgenic progestin, hormonal coil (IUS), the hormonal contraceptive implant or the DMPA hormonal injection;
2. History of DMPA hormonal injection use in those women not currently using the DMPA hormonal injection;
3. Diagnosed Premature Ovarian Insufficiency;
4. Pregnancy;
5. Less than 2 years postpartum;
6. Given birth to more than 2 children;
7. Evidence of disordered eating (≥ 20 on the EAT-26);
8. Any self-diagnosed eating disorder;
9. Self-reported change in body mass of ≥ 5% over the previous 3 months;
10. Body mass index of < 18 or > 30 kg·m2;
11. Evidence of menstrual disturbance (oligomenorrhea: < 9 menstrual cycles in previous 12 months or amenorrhoea: ≤ 3 menstrual cycles in the previous 12 months);
12. Habitual smoking (regularly smoking more than 10 cigarettes per day);
13. Taking any medications known to affect bone or calcium metabolism (e.g., treatment for thyroid disorders).
14. Total 25-hydroxyvitamin D (25(OH)D)level < 30 nmol/l at baseline, confirmed with a venous blood sample;
15. Self-declared history of heart, liver or kidney disease, diabetes, or thyroid disorder;
16. Self-reported bone fracture in the previous 12 months.

Exclusion Criteria for Reference Point Indentation Only:

1. Local oedema;
2. Local skin infection or cellulitis;
3. Prior clinical or stress fracture in the tibial diaphysis;
4. Dermatological lesions around the measurement site;
5. Focal tibial lesions like in primary or metastatic tumour, Paget's disease, Gaucher;
6. Osteomyelitis of the tibia;
7. Systemic infection or fever (unless unrelated to infection);
8. Allergy to lidocaine.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women of reproductive age.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Calcium balance. | Baseline measurement for long acting reversible contraceptive users. Day 21 and 28 of the pill cycle for the combined oral contraceptive pill users. Menses (day 0), mid-follicular, ovulation, and mid-luteal phase for non-users.
  The ratio of the calcium isotopes 44Ca:42Ca in first morning void urine.

SECONDARY OUTCOMES:
Circulating concentrations of reproductive hormones at rest following an overnight fast. | Baseline measurement for long acting reversible contraceptive users. Day 21 and 28 of the pill cycle for the combined oral contraceptive pill users. Menses (day 0), mid-follicular, ovulation, and mid-luteal phase for non-users.
  Fasted circulating concentration of luteinising hormone, follicle stimulating hormone, oestradiol, progesterone, testosterone, sex-hormone binding globulin.
Circulating concentrations of metabolic hormones at rest following an overnight fast. | Baseline measurement for long acting reversible contraceptive users. Day 21 and 28 of the pill cycle for the combined oral contraceptive pill users. Menses (day 0), mid-follicular, ovulation, and mid-luteal phase for non-users.
  Fasted circulating concentration of cortisol, cortisol binding globulin, insulin-like growth factor-1 (IGF-1), IGF binding protein 1, IGF binding protein 3, prolactin, relaxin, dehydroepiandrosterone sulfate, thyroid stimulating hormone, free thyroxine, free triiodothyronine.
Circulating concentrations of bone turnover markers at rest following an overnight fast. | Baseline measurement for long acting reversible contraceptive users. Day 21 and 28 of the pill cycle for the combined oral contraceptive pill users. Menses (day 0), mid-follicular, ovulation, and mid-luteal phase for non-users.
  Fasted circulating concentration of procollagen type 1 N-terminal propeptide (P1NP), bone specific alkaline phosphatase (bone ALP), beta carboxy-terminal cross-linking telopeptide of type 1 collagen (βCTX), intact parathyroid hormone, osteoprotegerin, receptor activator of nuclear factor kappa B ligand (RANKL), ionised and albumin-adjusted calcium, and phosphate.
Circulating concentrations of markers of resting iron status following an overnight fast. | Baseline measurement for long acting reversible contraceptive users. Day 21 and 28 of the pill cycle for the combined oral contraceptive pill users. Menses (day 0), mid-follicular, ovulation, and mid-luteal phase for non-users.
  Fasted circulating concentration of hepcidin-25, ferritin, soluble transferrin receptor, haemoglobin, and haematocrit.
Areal bone mineral density. | Single measurement at baseline for long acting reversible contraceptive users, day 21 for combined oral contraceptive users and at ovulation for non-users.
  Whole-body, lumbar spine, and neck of femur bone mineral density measured by dual-energy x-ray absorptiometry (DXA) scan.
Volumetric bone mineral density at the tibia and radius. | Single measurement at baseline for long acting reversible contraceptive users, day 21 for combined oral contraceptive users and at ovulation for non-users
  Tibial (4% and 30% site) and radial volumetric bone mineral density measured by high-resolution peripheral quantitative computed tomography.
Microarchitecture and structure at the tibia and radius. | Single measurement at baseline for long acting reversible contraceptive users, day 21 for combined oral contraceptive users and at ovulation for non-users
  Tibial (4% and 30% site) and radial microarchitecture, and geometry measured by high-resolution peripheral quantitative computed tomography.
Tibial bone material properties and strength | Single measurement for all groups taken no more than one month after completion of the study period.
  Tibial bone strength measured by reference point indentation.
Muscle function. | Baseline measurement for long acting reversible contraceptive users. Day 21 and 28 of the pill cycle for the combined oral contraceptive pill users. Menses (day 0), mid-follicular, ovulation, and mid-luteal phase for non-users.
  Isometric single-leg testing consisting of three maximal isometric contractions at 90° of knee flexion. Dynamic single-leg testing consisting of six repetitions at 60°/s, followed by 15 repetitions at 180°/s. Single-leg drop on each leg from a raised platform.
Muscle and tendon properties. | Baseline measurement for long acting reversible contraceptive users. Day 21 and 28 of the pill cycle for the combined oral contraceptive pill users. Menses (day 0), mid-follicular, ovulation, and mid-luteal phase for non-users.
  Digital palpation measurement of tone (Hz), stiffness (N/m) and elasticity of the rectus femoris, gastrocnemius, soleus, patella tendon and Achilles tendon using the Myoton device.

OTHER OUTCOMES:
Agreement between wearable detection of ovulation and ovulation inferred from luteinising hormone surge tests. | For one month prior to the start of the study period, and during the entire study period
  Urinary luteinising hormone surge test and menstrual cycle tracking using the commercially available Ava Bracelet.
Agreement between dual-energy x-ray absorptiometry and Echolight ultrasound bone mineral density. | Single measurement at baseline for long acting reversible contraceptive users, day 21 for combined oral contraceptive users, and at ovulation for non-users
  Bone mineral density of the lumbar spine and neck of femur, measured by dual-energy x-ray absorptiometry and Echolight ultrasound.
Body composition. | Single measurement at baseline for long acting reversible contraceptive users, day 21 for combined oral contraceptive users, and at ovulation for non-users
  Body mass, lean mass, and fat mass measured by dual energy x-ray absorptiometry.
Circulating concentrations of markers of vitamin D at rest. | Single measurement for all groups at pre-study visit.
  Fasted circulating concentration of total 25-hydroxyvitamin D (25(OH)D), free total vitamin D (25(OH)D), total 24,25 dihydroxyvitamin D, 1,25 dihydroxyvitamin D, and vitamin D binding protein.

CONTACTS AND LOCATIONS:
Locations (1):
- Army Health and Performance Laboratory, Camberley, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared pending approval from the UK Ministry of Defence.

REFERENCES:
- [Derived] Myers SJ, Knight RL, Wardle SL, Waldock KA, O'Leary TJ, Jones RK, Muckelt PE, Eisenhauer A, Tang JC, Fraser WD, Greeves JP. Effect of Menstrual Cycle and Hormonal Contraception on Musculoskeletal Health and Performance: Protocol for a Prospective Cohort Design and Cross-Sectional Comparison. JMIR Res Protoc. 2024 Jul 11;13:e50542. doi: 10.2196/50542. PMID 38990638